CLINICAL TRIAL: NCT05292105
Title: NC Xperience Post-Market Clinical Follow-up Study
Brief Title: NC Xperience PMCF Study( rEPIC04B)
Acronym: rEPIC04B
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: NC Xperience PMCF Study
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Coronary balloon dilatation catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: NC Xperience

INTERVENTIONS:
Device: NC Xperience — Coronary dilatation balloon catheter (non compliant)

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of NC Xperience to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with NC Xperience .

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the NC Xperience in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with NC Xperience according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

* Not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with NC Xperience according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 7 days
  Freedom from composite of cardiac death, myocardial infarction (MI) and Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Efficacy Endpoint. freedom from Target Lesion Failure | 7 days
  Freedom from composite of cardiac death, myocardial infarction (MI)and new Target Lesion Revascularization (TLR)
Freedom from Balloon rupture | During percutaneous coronary intervention (PCI)
  Freedom from Balloon rupture
Freedom from Hypotube rupture | During PCI
  Freedom from Hypotube rupture
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario Marques de Valdecilla, Santander

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Brodie BR, Cooper C, Jones M, Fitzgerald P, Cummins F; Postdilatation Clinical Compartative Study (POSTIT) Investigators. Is adjunctive balloon postdilatation necessary after coronary stent deployment? Final results from the POSTIT trial. Catheter Cardiovasc Interv. 2003 Jun;59(2):184-92. doi: 10.1002/ccd.10474. PMID 12772236
- [Background] Chandrasekhar J, Allada C, O'Connor S, Rahman M, Shadbolt B, Farshid A. Efficacy of non-compliant balloon post-dilation in optimization of contemporary stents: A digital stent enhancement study. Int J Cardiol Heart Vessel. 2014 Mar 19;3:43-48. doi: 10.1016/j.ijchv.2014.03.006. eCollection 2014 Jun. PMID 29450169
- [Background] Pasceri V, Pelliccia F, Pristipino C, Roncella A, Irini D, Varveri A, Bisciglia A, Speciale G. Clinical effects of routine postdilatation of drug-eluting stents. Catheter Cardiovasc Interv. 2014 May 1;83(6):898-904. doi: 10.1002/ccd.24999. Epub 2013 Dec 18. PMID 23703842
- [Background] Rana O, Shah NC, Wilson S, Swallow R, O'Kane P, Levy T. The impact of routine and intravascular ultrasound-guided high-pressure postdilatation after drug-eluting stent deployment: the STent OPtimization (STOP) study. J Invasive Cardiol. 2014 Dec;26(12):640-6. PMID 25480993
- [Background] Kim BG, Cho SW, Kim DH, Kim JH, Byun YS, Goh CW, Rhee KJ, Lee BK, Kim BO. Stent length is a contributing factor of suboptimal stent expansion in drug-eluting stents. Kardiol Pol. 2015;73(8):598-605. doi: 10.5603/KP.a2015.0034. Epub 2015 Mar 3. PMID 25733175